CLINICAL TRIAL: NCT04974528
Title: INHALE-1: A 26-week Primary Treatment Phase, With 26-week Extension, Open-label, Randomized Clinical Trial Evaluating the Efficacy and Safety of Afrezza® Versus Rapid-acting Insulin Analog Injections, Both in Combination With a Basal Insulin, in Pediatric Subjects With Type 1 or Type 2 Diabetes Mellitus
Brief Title: Afrezza® INHALE-1 Study in Pediatrics
Acronym: INHALE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-155 Part 2
Record Dates: First submitted 2021-06-22; First posted 2021-07-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Insulin; Inhaled; Afrezza; Technosphere; Pediatric
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Respiratory Aspiration | interventions — Insulin; Insulin, Short-Acting; Insulin Aspart; Insulin Lispro; insulin glulisine; Insulin Glargine; insulin degludec; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afrezza (Technosphere Insulin) + Basal Insulin (Experimental): Individualized dose of Afrezza (Technosphere Insulin) for each patient before each meal (breakfast, lunch, and dinner) for 26 weeks.
  Individualized basal insulin (insulin degludec, insulin glargine or insulin detemir) for each patient.
  Interventions: Biological: Afrezza; Biological: Basal Insulin
- RAA Injection + Basal Insulin (Active Comparator): Individualized dose of RAA injection (insulin aspart, insulin lispro or insulin glulisine) for each patient for 26 weeks.
  Individualized basal insulin (insulin degludec, insulin glargine or insulin detemir) for each patient.
  Interventions: Biological: Rapid-acting Insulin Analog; Biological: Basal Insulin

INTERVENTIONS:
Biological: Afrezza — Pharmaceutical form: powder
  Route of administration: inhalation
  Other Names: Technosphere Insulin
  Arms: Afrezza (Technosphere Insulin) + Basal Insulin
Biological: Rapid-acting Insulin Analog — Pharmaceutical form: clear and colorless solution for injection
  Route of administration: subcutaneous
  Other Names: insulin aspart; insulin lispro; insulin glulisine; Novolog®; Fiasp®; Humalog®; Admelog®; Apidra®
  Arms: RAA Injection + Basal Insulin
Biological: Basal Insulin — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: insulin glargine; insulin degludec; insulin detemir; Lantus®; Abasaglar®; Basaglar®; Semglee®; Toujeo®; Tresiba®; Levemir®

SUMMARY:
INHALE-1 is a Phase 3, open-label, randomized clinical study evaluating the efficacy and safety of Afrezza in combination with a basal insulin (i.e., the Afrezza group) versus insulin aspart, insulin lispro or insulin glulisine in combination with a basal insulin (i.e., the Rapid-acting Insulin Analog [RAA] injection group) in pediatric subjects with type 1 or type 2 diabetes mellitus. Following 26 weeks of randomized treatment (i.e., Afrezza or RAA injection combined with a basal insulin), all subjects will enter a treatment extension where subjects will receive Afrezza until Week 52. The purpose of the treatment extension is to assess safety and efficacy with continued use of Afrezza.

Pediatric subjects ≥4 and <18 years of age will be enrolled in this study. Subjects will be randomly assigned in a 1:1 ratio to either the Afrezza group or the RAA injection group.

The study is composed of:

* Up to 5-week screening/run-in period
* 26 week randomized treatment period
* 26-week treatment extension
* 4-week follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Assent from the pediatric subject, as appropriate, and fully informed consent from the parent(s) or legal guardian, as required by both state and federal laws and the local Institutional Review Board (IRB)
* Subjects ≥4 and <18 years of age
* Clinical diagnosis of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) per the Investigator and have been using insulin for at least 6 months for T1DM, or at least 3 months for T2DM
* Treatment with basal-bolus insulin therapy delivered by multiple daily injections for at least 2 weeks
* Bolus insulins are restricted to the RAAs insulin lispro, insulin aspart or insulin glulisine, including biosimilar products
* Basal insulins are restricted to insulin glargine, insulin degludec or insulin detemir, including biosimilar products
* Access to stable WiFi connection
* HbA1c ≥7.0% and ≤11%
* Average prandial dose of insulin ≥2 units per meal
* Utilized CGM for ≥70% of the time over a consecutive 14-day period preceding randomization

Exclusion Criteria:

* History of recent blood transfusions (within previous 3 months), hemoglobinopathies, or any other conditions that affect HbA1c measurements
* Recent history of asthma (defined as using any medications to treat within the last year), any other clinically important pulmonary disease (e.g., cystic fibrosis or bronchopulmonary dysplasia), or significant congenital or acquired cardiopulmonary disease
* History of serious complications of diabetes (e.g., active proliferative retinopathy or symptomatic autonomic neuropathy), or likely need for specific treatment for diabetic retinopathy (laser photocoagulation, vitrectomy, other) in the next year
* FEV1 and FEV1/forced vital capacity (FVC) ≤80% of predicted Global Lung Function Initiative (GLI) value
* Inability to achieve an acceptable FEV1 and FVC reading for subjects ≥8 years of age would make the subject ineligible
* For subjects <8 years of age who are unable to achieve an acceptable FVC reading, FEV1 only may be assessed; inability to achieve an acceptable FEV1 would make the subject ineligible
* Respiratory tract infection within 14 days before screening (subject may return 14 days after resolution of symptoms for rescreening)
* Inability or unwillingness to perform study procedures
* Exposure to any investigational product(s), including drugs or devices, in the past 30 days
* Any disease other than diabetes or exposure to any medication that, in the judgment of the Investigator, may impact glucose metabolism and current or anticipated acute uses of glucocorticoids or weight loss medications, with the exception of metformin and/or GLP-1 agonists (if GLP-1 agonists used for at least the 3 months prior to enrollment) in subjects with T2DM
* Use of antiadrenergic drugs (e.g., clonidine)
* Any concurrent illness (other than diabetes mellitus) not controlled by a stable therapeutic regimen
* Current uncontrolled eating disorder (e.g., anorexia or bulimia nervosa)
* Current drug or alcohol abuse or a history of drug or alcohol abuse that, in the opinion of the Investigator or the Sponsor, would make the subject an unsuitable candidate for participation in the study
* Smoking (includes cigarettes, cigars, pipes, marijuana, and vaping devices) for the preceding 6 months and/or positive urine cotinine test
* Female subject who is pregnant, breast-feeding, intends to become pregnant, or is of child-bearing potential, sexually active and not using adequate contraceptive methods as required by local regulation or practice
* An event of severe hypoglycemia, as judged by the Investigator, within the last 90 days prior to screening
* An episode of DKA requiring hospitalization within the last 90 days prior to screening

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 319 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 26 weeks
  Change in HbA1c from baseline to Week 26, for noninferiority assessment

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) | 26 weeks
  Change in FPG from baseline to Week 26, for superiority assessment
Event rate of pooled level 2 and level 3 hypoglycemia | 26 weeks
  Event rate of pooled level 2 and level 3 hypoglycemia (SMBG < 54 mg/dL and/or severe hypoglycemic events reported on the adverse event CRF) during the 26 -week randomized treatment period, for superiority assessment.
Change in HbA1c | 26 weeks
  Change in HbA1c from baseline to Week 26, for superiority assessment

OTHER OUTCOMES:
Event rate of level 1 hypoglycemia (SMBG <70 mg/dL) | 26 weeks
  Event rate of level 1 hypoglycemia during the 26-week randomized treatment period
Change in percent Time In Range (glucose 70 - 180 mg/dL) | 26 weeks
  Change in percent Time In Range from baseline to Week 26, using Continuous Glucose Monitoring (CGM)-derived data collected over the preceding 30 days for the 24-hour, daytime and nocturnal time periods
Change in percent time with glucose <54 mg/dL | 26 weeks
  Change in percent time with glucose <54 mg/dL from baseline to Week 26, using CGM-derived data collected over the preceding 30 days for the 24-hour, daytime and nocturnal time periods
Change in percent Time Below Range (glucose <70 mg/dL) | 26 weeks
  Change in percent Time Below Range from baseline to Week 26, using CGM-derived data collected over the preceding 30 days for the 24-hour, daytime and nocturnal time periods
Change in percent Time Above Range (glucose >180 mg/dL) | 26 weeks
  Change in percent Time Above Range from baseline to Week 26, using CGM-derived data collected over the preceding 30 days for the 24-hour, daytime and nocturnal time periods
Percentage of subjects with HbA1c <7.0% | At Week 26
  Percentage of subjects with HbA1c <7.0% at Week 26
Score of Diabetes Treatment Satisfaction Questionnaire (DTSQ) Change (c)-Teen | At Week 26
  Score of DTSQ(c)-Teen at Week 26 in the Afrezza group (score ranges from -24 to 24, with higher score means greater satisfaction)
Score of Diabetes Treatment Satisfaction Questionnaire (DTSQ) Change (c)-Parent | At Week 26
  Score of DTSQ(c)-Parent at Week 26 in the Afrezza group (score ranges from -30 to 30, with higher score means greater satisfaction)
Change in scores of DTSQ Status (s)-Teen | 26 weeks
  Change in scores of DTSQ(s)-Teen from baseline to Week 26 (change in score ranges from -48 to 48, with higher score means greater satisfaction)
Change in scores of DTSQ Status (s)-Parent | 26 weeks
  Change in scores of DTSQ(s)-Parent from baseline to Week 26 (change in scores ranges from -60 to 60, with higher score means greater satisfaction)
Change in HbA1c | 52 weeks (and 26 weeks if required)
  Change in HbA1c from baseline to Week 52 (and change from Week 26 to Week 52 if required) in subjects who switch from treatment with RAA injections to Afrezza at Week 26
Change in FPG | 52 weeks (and 26 weeks if required)
  Change in FPG from baseline to Week 52 (and change from Week 26 to Week 52 if required) in subjects who switch from treatment with RAA injections to Afrezza at Week 26
Change in percent Time In Range, Time Below Range and Time Above Range | 52 weeks (and 26 weeks if required)
  Change in percent Time In Range, Time Below Range and Time Above Range from baseline to Week 52 (and change from Week 26 to Week 52 if required) in subjects who switch from treatment with RAA injections to Afrezza at Week 26; using CGM-derived data collected over the preceding 30 days for the 24-hour, daytime, and nocturnal periods
Change in HbA1c | 52 weeks
  Change in HbA1c from baseline to Week 52 in subjects who receive Afrezza in both the randomized treatment period and the treatment extension
Change in FPG | 52 weeks
  Change in FPG from baseline to Week 52 in subjects who receive Afrezza in both the randomized treatment period and the treatment extension
Change in percent Time In Range, Time Below Range and Time Above Range | 52 weeks
  Change in percent Time In Range, Time Below Range and Time Above Range from baseline to Week 52 in subjects who receive Afrezza in both the randomized treatment period and the treatment extension; using CGM-derived data collected over the preceding 30 days for the 24-hour, daytime, and nocturnal periods
Score of DTSQ(c)-Teen at Week 52 | At Week 52
  Score of DTSQ(c)-Teen at Week 52 (after 6 months of Afrezza treatment) in subjects who switch from RAA injections to Afrezza (score ranges from -24 to 24, with higher score means greater satisfaction)
Score of DTSQ(c)-Parent at Week 52 | At Week 52
  Score of DTSQ(c)-Parent at Week 52 (after 6 months of Afrezza treatment) in subjects who switch from RAA injections to Afrezza (score ranges from -30 to 30, with higher score means greater satisfaction)
Change in scores of DTSQ(s)-Teen | 52 weeks
  Change in scores of DTSQ(s)-Teen from baseline to Week 52 (changes in score ranges from -48 to 48, with higher score means greater satisfaction)
Change in scores of DTSQ(s)-Parent | 52 weeks
  Change in scores of DTSQ(s)-Parent from baseline to Week 52 (change in scores ranges from -60 to 60, with higher score means greater satisfaction)
Event rates of hypoglycemic events | 52 weeks
  Event rates and incidence of total, nocturnal, and severe hypoglycemic events from baseline to Week 52
Incidence of hypoglycemic events | 52 weeks
  Incidence of total, nocturnal, and severe hypoglycemic events from baseline to Week 52
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 52 weeks
  Incidence and severity of TEAEs and SAEs from baseline to Week 52
Incidence and severity of Adverse Events of Special Interest (AESIs) | 52 weeks
  Incidence and severity of AESIs (i.e., acute bronchospasm, clinically relevant decline in pulmonary function [>15% decline from baseline percent predicted FEV1 accompanied by respiratory symptoms], hypersensitivity reactions [including anaphylaxis], use of asthma reliever medication, initiation or use of asthma controller medication, use of corticosteroid bursts, asthma exacerbations, hospitalization for asthma exacerbation, events of level 3 hypoglycemia, and diabetic ketoacidosis [DKA]) as well as the number of subjects with AESIs and number of individual events
Change in percent predicted Forced Expiratory Volume in 1 Second (FEV1) | 56 weeks
  Change from baseline to Weeks 13, 26, 39, 52, and 56 in percent predicted FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kaiserman, Study Director — Mannkind Corporation
Locations (39):
- United States (39):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Sutter Institute for Medical Research (formerly Center of Excellence in Diabetes and Endocrinology), Sacramento, California
  - University of California San Diego, Rady Children's Hospital, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Advent Health Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Iowa Diabetes Research, IDR, West Des Moines, Iowa
  - University of Louisville, Norton Children's Hospital, Louisville, Kentucky
  - Dr. Barry J. Reiner, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Michigan Pediatric Endocrine and Diabetes Services, Livonia, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - The DOCS, Las Vegas, Nevada
  - Atlantic Health, Morristown, New Jersey
  - UBMD Pediatrics Buffalo, Buffalo, New York
  - NYU Langone, Hassenfeld Children's Hospital, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oklahoma Children's Hospital, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - UT Southwestern, Dallas, Texas
  - DHR Health, Edinburg, Texas
  - Diabetes & Glandular Disease Clinic, DGD, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin